CLINICAL TRIAL: NCT00004198
Title: A Phase II Trial to Evaluate the Rate of Immune Response Using Idiotype Immunotherapies Produced by Molecular Biological Means for Treatment of Indolent B Cell Lymphoma
Brief Title: Vaccine Therapy Plus Sargramostim Following Chemotherapy in Treating Stage III or Stage IV Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genitope Corporation (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 0196-99-FB; P30CA036727 (NIH); GENITOPE-9901 (Other Grant/Funding Number: Genitope Corporation)
Record Dates: First submitted 2000-01-21; First posted 2004-05-21 (Estimated); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — keyhole-limpet hemocyanin; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Biological: keyhole limpet hemocyanin
Biological: sargramostim
Biological: tumor cell-based vaccine therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Vaccines may make the body build an immune response to kill tumor cells. Sargramostim may stimulate a person's immune system and help to kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of vaccine therapy plus sargramostim following chemotherapy in treating patients who have stage III or stage IV non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the ability of recombinant idiotype immunotherapy to stimulate a specific immune response against the B cell idiotype of the malignant clone that constitutes the tumor in patients with previously untreated stage III or IV indolent non-Hodgkin's lymphoma. II. Determine the safety and toxicity of this treatment regimen using Genitope Corporation's molecular rescue technology in this patient population.

OUTLINE: Patients receive induction chemotherapy consisting of oral cyclophosphamide, vincristine, and prednisone (CVP). Treatment repeats every 3 weeks until the maximal clinical response is achieved followed by 2 additional courses of consolidation therapy for up to a maximum of 10 courses. Patients not achieving adequate response receive up to 6 courses of alternate chemotherapy consisting of cyclophosphamide, doxorubicin, vincristine, and prednisone. At 3 months or up to 1 year following completion of chemotherapy, patients achieving adequate disease response receive vaccination consisting of recombinant tumor derived immunoglobulin idiotype with keyhole limpet hemocyanin conjugate subcutaneously (SQ) at 2 sites immediately followed by sargramostim (GM-CSF) SQ on day 1. Patients receive GM-CSF alone on days 2-4. Vaccination repeats every 4 weeks for 4 doses, followed 12 weeks later by the fifth and final dose. Patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage III or IV, indolent non-Hodgkin's lymphoma
* Follicular small cleaved cell
* Follicular mixed small cleaved and large cell with less than 50% large cells
* Tumor sample safely accessible by biopsy, needle aspiration, or phlebotomy
* Must have adequate circulating lymphoma cells
* Over 18 years old
* Karnofsky 80-100%
* WBC greater than 2,500/mm3
* Platelet count greater than 100,000/mm3
* Hemoglobin at least 10 g/dL
* Bilirubin less than 2 mg/dL
* SGOT/SGPT less than 2 times normal
* Creatinine less than 2 mg/dL
* HIV negative
* At least 2 months since prior non-physiologic doses of prednisone of greater than 20 mg or equivalent

Exclusion Criteria:

* No intermediate, high grade, or other non-Hodgkin's lymphomas (e.g., mantle cell, monocytoid B cell, marginal zone, small lymphocytic, chronic lymphocytic leukemia, or follicular large cell)
* No CNS metastasis
* No other illness or condition, including innate or pharmacologic immunosuppression, that would preclude study
* No other malignancy within the last 5 years except adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* No prior biologic therapy for lymphoma
* No prior cytotoxic therapy for lymphoma
* No prior steroids for lymphoma
* No concurrent maintenance steroids or greater than 5 mg of daily prednisone or equivalent
* No prior radiotherapy for lymphoma A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-06-25 (Actual); Primary Completion 2002-01-01 (Actual); Study Completion 2003-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie M. Vose, MD, Study Chair — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States